CLINICAL TRIAL: NCT04846569
Title: Adherence to HIV Treatment Postpartum: The Implications of Transitions Among Women Living With HIV in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: University of Cape Town (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1707001841; K01MH112443 (NIH)
Record Dates: First submitted 2021-04-08; First posted 2021-04-15 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: HIV; Pregnancy Related
Keywords: HIV; Pregnancy; Postpartum; South Africa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transition Theory-based Intervention (Experimental): Participants in the intervention arm will receive the Transition Theory-based intervention consisting of 4 sessions with a community health worker (2 during pregnancy, 2 postpartum) to support their transition from pregnancy to postpartum.
  Interventions: Behavioral: Transition Theory-based Intervention
- Enhanced Standard of Care Control (Active Comparator): Participants in the control arm will receive the standard of care plus one session with a community health worker.
  Interventions: Behavioral: Enhanced Standard of Care Control

INTERVENTIONS:
Behavioral: Transition Theory-based Intervention — The behavioral intervention is a theoretically driven curriculum focused on supporting mothers from pregnancy through postpartum in order to promote sustained HIV treatment adherence. Sessions utilize motivational interviewing and consist of a range of topics including motherhood, preparing for baby, disclosure, HIV education, adherence, birth experiences, support systems, and living positively.
  Arms: Transition Theory-based Intervention
Behavioral: Enhanced Standard of Care Control — In addition to standard of care, participants receive the first session of the Transition Theory-based Intervention curriculum which focuses on motherhood and preparation for baby but does not discuss the transition from pregnancy to postpartum or the postpartum period.
  Arms: Enhanced Standard of Care Control

SUMMARY:
Despite high levels of adherence motivation during pregnancy, HIV treatment adherence and engagement in care is difficult for women in the postpartum period. Supporting women during the transition from pregnancy to postpartum is imperative to sustaining HIV treatment adherence during this period. The investigators are conducting a small scale pilot study of a behavioral Transition Theory-based intervention to support ART adherence and engagement in ART services among pregnant and postpartum women living with HIV.

DETAILED DESCRIPTION:
Prevention of mother-to-child transmission (PMTCT) efforts have reduced the rates of vertical transmission to 2.7%, however, optimal antiretroviral therapy (ART) adherence remains a difficult goal to reach, particularly postpartum. Longitudinal qualitative research reveals a variety of facilitators and barriers to the transition from pregnancy to postpartum including employment/financial concerns, logistical concerns around childcare and breastfeeding, worries about vertical transmission and difficulties bonding. This intervention draws on the growing cadre of community health workers within the South African health care system and Transition Theory to develop a behavioral intervention to support women living with HIV through the transition from pregnancy to postpartum. The investigators are conducting a small scale pilot study to compare the impact of a Transition Theory-based intervention to enhanced standard of care on self-reported ART adherence and engagement in ART services among pregnant and postpartum women living with HIV.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. HIV positive status (based on clinic records)
3. Confirmed pregnant (based on clinic records) and estimated to be 23-34 weeks gestation (clinic records or self-report)
4. Currently prescribed ART
5. Planning on remaining a resident of Cape Town for at least 6 months postpartum
6. Ability to speak isiXhosa or English
7. Able to provide informed consent

Exclusion Criteria:

* Failure to meet any of the inclusion criteria
* Significant pre-existing psychiatric comorbidity at enrolment that may impact ability to consent according to the judgement of study personnel (including cognitive impairment or known psychotic disorder) Note: mothers will not be withdrawn from the study following foetal complications or death

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — We will enroll only pregnant women.
Enrollment: 62 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Pellowski, PhD, Principal Investigator — Brown University
Locations (1):
- Gugulethu Community Health Centre, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets will be made available by request, subject to agreement to Access Criteria, see below
Supporting Information: Study Protocol, ICF
Time Frame: After primary data has been published (anticipated September 2022), by request
Access Criteria: (1) a commitment to use the data only for research purposes and not to identify any individual participant; (2) a commitment to secure the data using appropriate computer technology and established security measures; (3) a plan for the dissemination of results; (4) appropriate authorship and recognition of all partners; and (5) a commitment to destroy or return the data after analyses are completed.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between April 2021 and March 2022 at the Gugulethu Midwife Obstetrics Unit (MOU), Cape Town, South Africa.
Pre-assignment Details: Participants completed consent on a separate day from baseline and randomization.
Period: Overall Study
Arm/Group | Transition Theory-based Intervention | Enhanced Standard of Care Control
Started | 23 | 20
Completed | 20 | 19
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transition Theory-based Intervention | Enhanced Standard of Care Control | Total
Number analyzed (Participants) | 23 | 20 | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33 (5.62) | 32 (6.13) | 33 (5.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 43
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black South African | 23 | 20 | 43
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 23 | 20 | 43
Baseline self-report ART Adherence [Mean (Standard Deviation); unit: units on a scale] — self-reported adherence using Wilson's 3 item adherence scale. Scores are transformed to follow a scale from 0-100 in which 100 is perfect adherence
  units on a scale | 80.72 (2.41) | 76.84 (2.09) | 78.92 (1.62)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the Intervention - Number of Counseling Sessions
Description: Feasibility will be assessed through the number of counseling sessions completed.
Time Frame: 3 months postpartum
Population: Transition Theory-based intervention participants received 4 counseling sessions compared to 1 session for those in the enhanced standard of care control condition; means are reported based on these denominators and should not be compared by condition
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | Transition Theory-based Intervention | Enhanced Standard of Care Control
Number analyzed (Participants) | 23 | 20
sessions | 2.92 (1.28) | 1 (0)

2. Primary Outcome: Preliminary Efficacy - ART Adherence
Description: Preliminary efficacy will be assessed as the correlation between study arm and self-reported HIV adherence on the 3 item Wilson ART adherence scale (self-report, 3 item scale recoded as 0-100, 100 indicating perfect adherence in the past month) at 6 months postpartum.
Time Frame: 6 months postpartum
Population: There was substantial LTFU for the 6 month postpartum timepoints. Analyses are conducted with all participants for whom these assessments were collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transition Theory-based Intervention | Enhanced Standard of Care Control
Number analyzed (Participants) | 11 | 13
score on a scale | 82.65 (11.15) | 82.73 (8.82)
Statistical Analysis 1: Comparison: Transition Theory-based Intervention vs Enhanced Standard of Care Control; Test type: Superiority; Mean Difference (Final Values) = 0.004, 95% CI 2-sided [-0.38 to 0.39]

3. Primary Outcome: Preliminary Efficacy- Retention in HIV Services
Description: Preliminary efficacy will be assessed as the correlation between study arm and retention in HIV services at 6 months postpartum. Retention in HIV services is measured by clinic records. Retention at 6 months postpartum is measured as attended HIV clinic appointment in the past 3 months.
Time Frame: 6 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Transition Theory-based Intervention | Enhanced Standard of Care Control
Number analyzed (Participants) | 20 | 19
Participants | 17 | 15
Statistical Analysis 1: Comparison: Transition Theory-based Intervention vs Enhanced Standard of Care Control; Test type: Superiority; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.78 to 0.47]

4. Primary Outcome: Preliminary Efficacy-viral Suppression
Description: Preliminary efficacy will be assessed as the correlation between study arm and viral suppression at 6 months postpartum. Viral suppression will be measured by clinic records, with viral suppression defined as HIV viral load less than 200 copies/mL.
Time Frame: 6 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Transition Theory-based Intervention | Enhanced Standard of Care Control
Number analyzed (Participants) | 11 | 7
Participants | 11 | 7
Statistical Analysis 1: Comparison: Transition Theory-based Intervention vs Enhanced Standard of Care Control; All participants who we were able to obtain records for were virally suppressed thus an effect size was unable to be calculated; Test type: Superiority; All participants who we were able to obtain records for were virally suppressed thus an effect size was unable to be calculated as originally planned

5. Secondary Outcome: Adherence Self-efficacy - Confidence in Taking Medications
Description: Adherence self-efficacy will be measured using the AACTG adherence self-efficacy scale, 15 items, using 5 point Likert scale ranging from not confident at all to very confident. Total scores range from 15-75, with higher scores indicating higher self-efficacy.
Time Frame: 6 months postpartum
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transition Theory-based Intervention | Enhanced Standard of Care Control
Number analyzed (Participants) | 14 | 11
units on a scale | 63.93 (4.95) | 69.55 (0.45)
Statistical Analysis 1: Comparison: Transition Theory-based Intervention vs Enhanced Standard of Care Control; Test type: Superiority; Median Difference (Final Values) = 0.20, 95% CI 2-sided [-0.20 to 0.53]

6. Secondary Outcome: Acceptability/Utility of the Intervention
Description: Acceptability of the Transition Theory-based intervention, assessed during in-depth interviews among participants in the intervention condition to gauge general feelings of acceptability and perceived usefulness of the intervention.
Time Frame: 6 months postpartum
Population: 11 participants randomized to the intervention arm completed qualitative interviews following the 6 month follow-up assessment and are used in the qualitative analysis. Count represents number of participants who reported positively about the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Transition Theory-based Intervention
Number analyzed (Participants) | 11
Participants | 11
Statistical Analysis 1: Comparison: Transition Theory-based Intervention; Test type: Other — Qualitative data analysis; Thematic qualitative data analysis was conducted to determine the count of participants reporting positively about the intervention

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Transition Theory-based Intervention | Enhanced Standard of Care Control
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/20
Other Adverse Events (participants affected / at risk) | 0/23 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT04846569/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT04846569/ICF_001.pdf